CLINICAL TRIAL: NCT03416296
Title: Evaluation of Role of Ultrasound TA,TV,TP in Diagnosis of Placenta Previa and MAP(Morbidly Adherent Placenta )
Brief Title: Role of Ultrasound in Diagnosis of Placenta Previa and MAP
Status: Completed | Type: Observational
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: placenta
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Morbidly Adherent Placenta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — uterus in case of hysterectomy after cesarean hysterectomy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal placenta: TA , TV ,TP us
- placenta previa and MAP: TA,TV.TP us

SUMMARY:
Placenta accreta occurs when the placental implantation is abnormal. The marked rise in incidence has been assumed the increasing prevalence of cesarean delivery in recent years.

DETAILED DESCRIPTION:
The most accepted theory is that abnormal placentation . The most important risk factor for placenta accreta is placenta previa after a prior cesarean delivery. The first clinical manifestation of placenta accreta is usually severe , life-threatening hemorrhage. The recommended intervention of suspected placenta accreta is planned preterm cesarean hysterectomy with the placenta left in situ.

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies with previous cesarean sections
* GA above 30 weeks

Exclusion Criteria:

* Primigravida patients
* GA below 30 weeks

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females with GA above 30 weeks
Study Population: pregnant females with previous cs will be subjected to US to assess placental location and MAP
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
number of participants who will be diagnosed to have normal placenta or placenta previa or morbidly adherent placenta by US | within 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt